CLINICAL TRIAL: NCT01609569
Title: Utility of Pro-calcitonin as an Indicator of Ischemia in Patients Undergoing Percutaneous Coronary Intervention With Subsequent Coronary Complications.
Brief Title: Pro-calcitonin Marker as Indicator of Ischemia in Patients With Complicated Coronary Intervention.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Saint Michael's Medical Center (Other)
Responsible Party: Principal Investigator, Habib Habib, MD, Principal Investigator, Saint Michael's Medical Center
Other Study IDs: #09/12
Record Dates: First submitted 2012-05-29; First posted 2012-06-01 (Estimated); Last update posted 2013-02-22 (Estimated); Status verified 2013-02

CONDITIONS: Coronary Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- coronary complication: patients with coronary complication and patients without coronary complications.
  pro-calcitonin will be measured in both groups to see if any correlation.

SUMMARY:
The aim of this study is to determine on preliminary basis weather an elevated pro-calcitonin level can be used to assess ischemia as a result of coronary artery complications during percutaneous coronary intervention (PCI).

DETAILED DESCRIPTION:
Pro-calcitonin is a type of protein found in the blood. This protein has recently be found to be elevated in patients with diseases of the arteries of the heart such as heart attack.

Percutaneous coronary intervention (PCI) is widely used in the treatment of many patients with blockage in the arteries of the heart.

the investigators normally used a marker called troponin after cardiac catheterization. However, this marker may not be specific.

Pro-calcitonin has been found to be a useful marker for the detection of myocardial injury. the value of Pro-calcitonin as a marker for the identification of myocardial damage undergoing PCI has not yet been studied.

ELIGIBILITY:
Inclusion Criteria:

* patients older than 18 years old.

Exclusion Criteria:

* no consent.
* suspicion of sepsis.
* Patients with elevated troponin or procalcitonin before enrollment.
* patients who had non-elective angioplasty (e.g. rescue angioplasty, primary angioplasty, salvage angioplasty, or emergency angioplasty)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-05; Primary Completion 2014-04 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Pro-calcitonin blood level | "0,24 hours post cardiac intervention"

CONTACTS AND LOCATIONS:
Overall Officials: Habib Habib, MD, Principal Investigator — Saint Michael's Medical Center; Fayez Shamoon, MD,FACC, Study Director — Saint Michael's Medical Center; yaser elnhar, MD, Study Chair — Saint Michael's Medical Center; Vincent Debari, PhD, Study Chair — Saint Michael's Medical Center; Ashraf Jmeian, MD, Study Chair — Saint Michael's Medical Center; Ahmad Isbitan, MD, Study Chair — Saint Michael's Medical Center
Locations (1):
- Saint Michael's Medical Center, Newark, New Jersey, United States

REFERENCES:
- [Background] Sinning CR, Sinning JM, Schulz A, Schnabel RB, Lubos E, Wild PS, Papassotiriou J, Bergmann A, Blankenberg S, Munzel T, Bickel C; AtheroGene Study Investigators. Association of serum procalcitonin with cardiovascular prognosis in coronary artery disease. Circ J. 2011;75(5):1184-91. doi: 10.1253/circj.cj-10-0638. Epub 2011 Mar 3. PMID 21378450